CLINICAL TRIAL: NCT05013359
Title: Awareness, Care & Treatment In Obesity Management - An International Observation Among Teens (ACTION Teens)
Acronym: ACTION Teens
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-003; U1111-1262-1190 (Other: World Health Organization)
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents Living with Obesity (ALwO): Recruited from online, general population consumer panels
  Interventions: Other: No treatment given
- Health Care Providers (HCPs): HCPs treating adolescents who have obesity
  Interventions: Other: No treatment given
- Caregivers: A parent or legal guardian of an adolescent with obesity
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
ACTION Teens is a multinational cross-sectional survey-based study. The study consists of a quantitative online survey to be conducted among three groups of respondents in ten countries worldwide. The respondent population will include Adolescents Living with Obesity (ALwO), Caregivers of ALwO, and HCPs treating adolescents who have obesity.

The goal of this study is to provide insights to drive awareness around the needs of adolescents living with obesity and their caregivers, as well as to identify key areas of misalignment between adolescents, their caregivers and the HCPs involved in obesity treatment and management. ACTION Teens is designed to generate evidence to identify and address these challenges on both a global and local level, extending the insights from the previously conducted ACTION-IO study.

ELIGIBILITY:
Inclusion Criteria for Adolescents living with obesity:

* Informed consent obtained by parent/legal guardian and ALwO before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, aged 12 to less than 18 years at the time of signing informed consent.
* Lives in one of the participating countries: Italy, Spain, UK, Mexico, Colombia, Australia, Saudi Arabia, Turkey, South Korea, and Taiwan.
* Has a current BMI-for-age (based on self-reported sex, age, height, and weight) greater than or equal to 95th percentile for age and sex based on charts appropriate locally for the country of residence.

Inclusion Criteria for Caregivers of Adolescents living with obesity:

* Informed consent before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 24 years at the time of signing informed consent.
* Lives in one of the participating countries: Italy, Spain, UK, Mexico, Colombia, Australia, Saudi Arabia, Turkey, South Korea, and Taiwan.
* Has an adolescent in the household with a current BMI-for-age (based on self-reported sex, age, height, and weight) greater than or equal to 95th percentile for age and sex based on charts appropriate locally for the country of residence.
* Resides in the same household as the ALwO at least 50% of the time.
* Is involved in the healthcare decisions of the ALwO.

Inclusion Criteria for Health Care Providers:

* Informed consent before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Is a physician.
* Practices in one of the participating countries: Italy, Spain, UK, Mexico, Colombia, Australia, Saudi Arabia, Turkey, South Korea, and Taiwan
* In clinical practice more than or equal to 2 years.
* Spends at least 50% of time in direct patient care.
* Has seen/treated at least ten adolescent patients (age 12 to less than 18 years) with obesity in a typical month (defined as BMI-for-age greater than or equal to 95th percentile for age and sex based on charts appropriate locally for the country of residence).

Exclusion Criteria for Adolescents living with obesity:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness, inability, or language barriers precluding adequate understanding or cooperation.
* Has had significant weight loss or weight gain due to major injury or illness/condition (e.g., cancer, accident, pregnancy) in the past 6 months.
* Considers themselves to be extremely muscular.

Exclusion Criteria for Caregivers of Adolescents living with obesity:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness, inability, or language barriers precluding adequate understanding or cooperation.
* ALwO they care for has had significant weight loss or weight gain due to major injury or illness/condition (e.g., cancer, accident, pregnancy) in the past 6 months.
* Considers the ALwO they care for to be extremely muscular.

Exclusion Criteria for Health Care Providers:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness, inability, or language barriers precluding adequate understanding or cooperation.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The respondent population will include Adolescents living with obesity (ALwO), Caregivers of ALwO, and HCPs treating adolescents who have obesity.
Sampling Method: Non-Probability Sample
Enrollment: 12987 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Attitudes about obesity, attitudes about people with obesity, and beliefs about the impact of obesity | At the time of survey response (Day 1)
  5-point Likert scales (e.g., agreement, impact, frequency)
  - Proportion of responses in each category will be reported.
Weight loss attempts in past year, motivations to lose weight, barriers to losing weight, and definition of successful weight loss/management | At the time of survey response (Day 1)
  Yes/No; percentage of participants
  Multi-select from defined list
  - Percentage of respondents selecting an item or items will be reported.
History and frequency of conversations about weight, initiator of weight conversations, and responsibility for initiating weight conversations that occur between adolescents living with obesity/their caregivers and healthcare providers | At the time of survey response (Day 1)
  Numeric entry; percentage of participants Single select from defined list; percentage of time each initiates Single select from defined list
Assessment of interactions between adolescents living with obesity/their caregivers and healthcare providers, reasons why obesity may not be discussed, frequency of obesity diagnosis, and frequency of follow-up appointments made to discuss obesity | At the time of survey response (Day 1)
  5-point Likert scales Multi-select from defined list Yes/No; percentage of patients Yes/No; percentage of patients
Sources of information used to learn about obesity, healthy lifestyles, weight loss, and weight management | At the time of survey response (Day 1)
  Multi-select from defined list

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (10):
- Novo Nordisk Investigational Site, Sydney, Australia
- Novo Nordisk Investigational Site, Bogotá, Colombia
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Mexico City, Mexico
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Gatwick, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Kwok C, Bentley N, Curran J, Lister N, Truby H, Baur LA. Misaligned Attitudes and Perceptions Among Adolescents Living With Obesity, Caregivers and Healthcare Professionals: ACTION Teens Australia Survey Study. J Paediatr Child Health. 2025 Oct;61(10):1573-1581. doi: 10.1111/jpc.70146. Epub 2025 Jul 14. PMID 40657891
- [Derived] Halford JCG, Brown A, Clare K, Ells LJ, Ghosh A, Giri D, Hughes C, Senniappan S. Insights from the ACTION Teens Study: a survey of adolescents living with obesity, their caregivers and healthcare professionals in the UK. BMJ Open. 2024 Jul 23;14(7):e086391. doi: 10.1136/bmjopen-2024-086391. PMID 39043586
- [Derived] Maffeis C, Busetto L, Wasniewska M, Di Pauli D, Maccora C, Lenzi A. Perceptions, attitudes, and behaviors among adolescents living with obesity, caregivers, and healthcare professionals in Italy: the ACTION Teens study. Eat Weight Disord. 2024 May 8;29(1):35. doi: 10.1007/s40519-024-01663-7. PMID 38717596
- [Derived] Mooney V, Baur LA, Bereket A, Bin-Abbas B, Chen W, Fernandez-Aranda F, Nieto NG, Lopez Siguero JP, Maffeis C, Osorto CK, Reynoso R, Rhie YJ, Toro-Ramos M, Halford JC. The views of teenagers with obesity, their caregivers, and doctors: a plain language summary of the ACTION Teens global survey. J Comp Eff Res. 2023 Jan;12(1):e220164. doi: 10.2217/cer-2022-0164. Epub 2022 Oct 20. PMID 36264113